CLINICAL TRIAL: NCT06089577
Title: Effects of Cangrelor on MIcRovAscular Disfunction During Elective Percutaneous CORonary Intervention
Acronym: MIRACOR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Luigi Di Serafino, Assistant Professor of Cardiology, MD, PhD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 373/2023
Record Dates: First submitted 2023-10-05; First posted 2023-10-18 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Coronary Artery Disease
Keywords: index of microcirculatory resistance; coronary flow reserve; Cangrelor
MeSH Terms: conditions — Coronary Artery Disease | interventions — cangrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cangrelor (Experimental): In the Experimental group, before performing PCI, all patients will be treated with Cangrelor (Kangrexal) with an i.v. loading bolus (30mg/Kg) followed by i.v. infusion (4mg/Kg/min) for 2 hours. At the end of the infusion, as per current clinical practice, a loading dose of Clopidogrel (600mg) will be administered. A manteinance daily dose of 75mg will be associated with oral ASA (100mg).
  Interventions: Drug: Cangrelor 50 MG
- Control (No Intervention): In the Control group, either before or after PCI a loading dose of Clopidogrel will be administered and a manteinance daily dose of 75mg will be associated with oral ASA (100mg). PCI procedure will be performed as per current cinical practice, according clinical guidelines and at operator discretion.

INTERVENTIONS:
Drug: Cangrelor 50 MG — Cangrelor will be administered during PCI
  Arms: Cangrelor

SUMMARY:
Dual Antiplatelet Therapy represents the main therapy for patients presenting with chronic coronary syndromes and undergoing elective PCI. However, most of these patients are not properly covered in terms of inhibition of platelets aggregation at the time of PCI, and are exposed to an higher risk of microvascular damage which in turns might be responsible of residual symptoms persistence and the findings of residual ischemia at the non-invasive tests. In naïve patients, cangrelor can be administered at the time of PCI potentially protecting coronary microcirculation. The aim of this randomized study is indeed to evaluate the use of Cangrelor as compared with standard practice (with Clopidogrel) in terms of incidence of coronary microvascular dysfunction following elective PCI of functionally significant intermediate coronary stenoses. All consecutive patients, fulfilling inclusion and exclusion criteria, will be enrolled and both FFR and CFR/IMR will be measured before and after PCI. Platelet reactivity will be also evaluated mainly during PCI procedure. At 30 days of follow up, patients will be interrogated about symptoms persistence and will be asked to complete the specific Seattle Angina Questionaty (SAQ7). At 3 months a SPECT could be performed in order to evaluate the presence of residual ischemic area in the myocardial territory downstream to the treated vessel. With this study we will be able to evaluate the potential benefit of using Cangrelor, as compared with standard therapy with Clopidogrel, in terms of protection of coronary microcirculation during elective PCI and reduction of both residual symptoms and ischemia at clinical follow up.

DETAILED DESCRIPTION:
Background and state of the art Dual antiplatelet therapy (DAPT) is the main therapy for patients presenting with chronic coronary syndrome (CCS) undergoing elective percutaneous coronary interventions (PCI). It is mainly represented by acetylsalicylic acid (ASA) and Adenosine-diphosphate (ADP) receptor antagonists, such as Clopidogrel, Prasugrel and Ticagrelor. However, pretreatment with DAPT in patients undergoing elective PCI is only considered optional, thereby a large proportion of these patients is not adequately treated at the moment of PCI.1, 2 Manipulations of the coronary arteries during PCI, particularly when complex procedures are performed, might favor platelets aggregation and small thrombus formations with distal embolization.3, 4 In addition, the higher platelet reactivity in this context is associated with endothelial dysfunction which might favour the higher incidence of microvascular damage during PCI.5-9 This latter might be responsible of persistence of angina symptoms even after successfull PCI.10-12 In the setting of CCS and elective PCI, ASA is mainly associated with Clopidogrel. This latter is an oral pro-drug which needs to be converted by the liver in an active metabolite which is able to inhibit the ADP receptor in few hours after the loading dose. However, some patients might be resistent to Clopidogrel with inadeguate platelets inhibition and higher risk of ischemic events.1, 2 Normally, in naïve patients, Clopidogrel is administered at the end of the procedure with an oral loading dose of 600mg, followed by 75mg per day, while ASA can be administered as soon as possible by endovenous bolus (250mg).

Cangrelor is an analogous of the ADP which inhibits platelets aggregation in few minutes after endovenous administration, thereby it can be administered at the moment of PCI potentially reducing the risk of microvascular damage as compared with regular practice.13 This drug is currently recommended by the European guidelines for coronary revascularization in CCS patients, not on treatment with other ADP receptor antagonists.

Objectives The main purpose of the present randomised and open-label study will be the comparison between Cangrelor and regular practice with Clopidogrel in terms of incidence of microvascular damage in CCS patients undergoing elective PCI. The assessment of microvascular damage will be performed by measuring the index of microvascular resistance (IMR) before and after PCI. Even though recommended by the current European guidelines, cangrelor has never been evaluated with the purpose to protect microcirculation during PCI and this study might highlight the potential benefit of Cangrelor, as compared with regural practice, in the context of elective PCI. In addition, as secondary objectives, the occurrence of peri-procedural myocardial infarction (MI) will be evaluated and platelets reactivity will be also assessed with the aim to correlate platelets reactivity with IMR values, supporting the correlation between platelets reactivity and endothelial dysfunction.

At 30 and 90 days of follow-up, patients will report on the persistence of angina symptoms by completing a specific questionary (SAQ7). This point is also of interest, since coronary microvascular dysfunction (IMR>25) might be responsible of angina symptoms regardless of the presence of epicardial stenosis. Microvascular dysfuction can be detected either before PCI or after PCI as result of microvascular damage. Although with poor prognostic value, microvascular damage might be responsible of persistence of typical symptoms and ischemic signs at non-invasive tests despite a successful PCI, leading patients towards the esecution of several and useless non-invasive and invasive tests. Thereby, the protection of the coronary microcirculation during elective PCI might significantly reduce the persistence of typical symptoms in post-PCI patients and finally provide a significant savings for the heath care system.

Methodology and work plan This will be a randomised and open-label study, including all consecutive patients presenting with chronic coronary syndromes not on treatment with any of the ADP receptor antagonists, and undergoing elective PCI of functionally significant intermediate de-novo coronary artery stenoses. Patients presenting with ACS or heart failure (left ventricle ejection fraction < 30%) will be excluded as well as patients with a subtotal occlusion of a major coronary artery not requiring FFR evaluation.

* Pre-procedural assessment. All patients will be screened before the procedure and will be asked to answer the specific angina questionary (Seattle Angina Questionnaire SAQ-7), for the assessment of the severity of the angina symptoms.
* Coronary angiography and functional assessment of intermediate coronary artery stenoses. Coronary angiography will be performed as per regular practice through the radial or femoral access in order to evaluate the presence of any epicardial stenoses in a major vessel. In this case, the ischemic potential of each stenosis will be assessed with the Fractional Flow Reserve (FFR), as also recommended by the current European guidelines.14, 16 Briefly, a pressure/temperature guidewire will be advanced beyond the stenosis and during i.v. adenosine induced maximal hyperemia the ratio between distal (Pd) and proximal (Pa) pressures will be calculated. A FFR value ≤ 0.80 will identify a functionally significant coronary stenosis with indication to perform PCI. With the same guidewire, and the same setting, it will be also possible to measure both the Coronary Flow Reserve (CFR) and the Index of Microcirculatory Resistance (IMR).17-19
* Randomization and PCI procedure. After the evaluation of both inclusions and exclusions criteria, patients will be randomised in a 1:1 allocation ratio in two groups: 1) Experimental Group 2) Control Group. RedCap software will be used to randomise and to manage patients data. In the Experimental group, before performing PCI, all patients will be treated with Cangrelor (Kangrexal) with an i.v. loading bolus (30mg/Kg) followed by i.v. infusion (4mg/Kg/min) for 2 hours. At the end of the infusion, as per current clinical practice, a loading dose of Clopidogrel (600mg) will be administered. A manteinance daily dose of 75mg will be associated with oral ASA (100mg). In the Control group, either before or after PCI a loading dose of Clopidogrel will be administered and a manteinance daily dose of 75mg will be associated with oral ASA (100mg). PCI procedure will be performed as per current cinical practice, according clinical guidelines and at operator discretion.14
* Assessment of Platelets reactivity (PR). Blood samples for platelet function analysis will be collected in the catheterization laboratory through the arterial sheath. PR will be measured with the VeryfyNow system in three different time points, without interfering with the regular PCI procedure:

  * Time 0: Before PCI and Cangrelor/Clopidogrel administration;
  * Time 1: At the end of the PCI procedure and within 1 hour from the administration of Cangrelor/Clopidogrel.
  * Time 2: At 4-6 hours from PCI procedure.
* Post PCI assessment. Both FFR and CFR/IMR will be assessed at the end of the PCI with the purpose to evaluate 1) the completeness of the revascularization from a functional standpoint and 2) the occurrence of microvascular damage. This latter will be diagnosed in case of Post-PCI IMR values > 25 if Pre-PCI IMR values are normal (<25) or, in case of abnormal Pre-PCI IMR values, if Post-PCI values will be 20% higher.
* Non-invasive Post-PCI assessment. Blood samples will be collected at 12 and 24 hours with the aim to evaluate the occurrence of peri-procedural MI defined as follow:

  * The finding of high sensitive Troponine I (hsTrop-I) values higher than 5X the ULN, in patients with normal hsTrop-I before PCI;
  * The finding of hsTrop-I values higher than 20% the baseline values, in patients with abnormal hsTrop-I before PCI;

In addition, the following criteria should also be fulfilled:

* ECG ischemic modification after PCI
* The findings of new Q waves at ECG
* The findings at the angiography of some modifications consistent with the hdTrop-I increase (i.e. side branch occlusion/dissection, distal embolization).

  * Follow-up. Patients will be followed up at 30 and 90 days. Besides clinical assessment, patients will be asked to complete SAQ7 questionary in order to evaluate the severity of residual symptoms, if any. In addition, at 90 days only, all patienst will perform a single photon emission computed tomography (SPECT) in order to evaluate the presence of ipoperfused areas downstream to the treated vessel.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients;
* Signed Informed Consent;
* Chronic coronary syndromes;
* P2Y12-inhibitors naive patients;
* Elective PCI of a functionally significant (FFR ≤ 0.80) de-novo intermediate coronary artery stenoses in a major vessel;

Exclusion Criteria:

* Underaged patients;
* Acute Conorary Syndromes;
* Already on treatment with P2Y12-inhibitors;
* Heart failure with severe reduction of the left ventricle ejection fraction (LVEF < 30%);
* Subtotal occlusion (diameter stenosis > 90%) of the target lesion;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of microvascular dysfunction | within 60 minutes post PCI procedures
  IMR > 25

SECONDARY OUTCOMES:
Periprocedural platelect reactivity | within 60 minutes post PCI procedures
  P2Y12 Reaction Units
Periprocedural platelect reactivity | within 180 minutes post PCI procedures
  P2Y12 Reaction Units
Incidence of Periprocedural myocardial infarction | within 24 hours post PCI procedures
  IV Universal Definition of Myocardial Infarction
Incidence of Residual Angina | 30 days post PCI
  SAQ7 questionnaire
Incidence of residual ischemia | 90 days post PCI
  SAQ7 questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Division of Cardiology, University Hospital of Ferrara, Ferrara
  - Division of Cardiology - Federico II University Hospital, Naples